CLINICAL TRIAL: NCT02061670
Title: A Multi-Centre, Double-Blind, Randomised, Placebo-Controlled Parallel-Group Study to Assess the Safety and Tolerability of Ragweed-SPIRE in Subjects With Asthma and Ragweed-Induced Rhinoconjunctivitis
Brief Title: Safety Study of Ragweed-SPIRE in Subjects With Ragweed Allergies and Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR007
Record Dates: First submitted 2014-02-03; First posted 2014-02-13 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Seasonal Allergic Rhinitis; Asthma
Keywords: Ragweed; Allergy; rhinoconjunctivitis; rhinitis; asthma
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Asthma; Hypersensitivity; Rhinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ragweed-SPIRE 1 (Experimental): Ragweed-SPIRE regimen 1 given 2 weeks apart
  Interventions: Biological: Ragweed-SPIRE
- Ragweed-SPIRE 2 (Experimental): Ragweed-SPIRE regimen 2 given 2 weeks apart
  Interventions: Biological: Ragweed-SPIRE
- Placebo (Placebo Comparator): Placebo given 2 weeks apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ragweed-SPIRE — Intradermal injection
  Arms: Ragweed-SPIRE 1; Ragweed-SPIRE 2
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether it is safe to administer Ragweed-SPIRE to subjects suffering from both ragweed allergy and asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years.
* Asthma treated by inhaled SABA or inhaled SABA plus low-medium dose ICS in 6 weeks prior to randomisation.
* A reliable history consistent with moderate to severe rhinoconjunctivitis on exposure to ragweed for at least the previous two ragweed seasons.
* Positive skin prick test to ragweed
* Ragweed-specific Immunoglobulin E (IgE) ≥ 0.35 kU/L.

Exclusion Criteria:

* History of life-threatening asthma.
* Uncontrolled asthma according to GINA
* FEV1 of < 70 % of predicted, regardless of the cause.
* Administration of adrenaline (epinephrine) is contraindicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* History of severe drug allergy or anaphylactic reaction to food.
* A history of any significant disease or disorder (e.g. immune system, pulmonary, cardiovascular, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment, history of alcohol or drug abuse)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Throughout subjects participation in the study, approximately 22 weeks

SECONDARY OUTCOMES:
Number of subjects with asthma exacerbations as a measure of safety and tolerability | Throughout subjects participation in the study, approximately 22 weeks
Evaluation of change in lung function as a measure of safety and tolerability | Throughout subjects participation in the study, approximately 22 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Kanata Allergy Services, Kanata, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Cheema Research Inc, Mississauga, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Inflamax Research, Toronto, Ontario